CLINICAL TRIAL: NCT06773793
Title: The Diagnostic Value of Shear Wave Elastography and Viscosity Imaging Techniques in Diabetic Peripheral Neuropathy
Status: Enrolling by invitation | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Dr. weijing zhang, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: NDTHNanjingUMS.
Record Dates: First submitted 2025-01-04; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Peripheral Neuropathy (DPN)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Observational controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The main objective of this observational study is to evaluate the diagnostic value of multimodal ultrasound for diabetic peripheral neuropathy (DPN). The questions it aims to address are: (1) To compare the differences in various parameters between the DPN group, non-DPN group, and healthy control group; (2) To explore the diagnostic efficacy of each parameter for DPN and establish a combined model.

ELIGIBILITY:
Inclusion Criteria:Individuals aged 18 to 75 years without diabetes -

Exclusion Criteria:Individuals without peripheral neuropathy.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinically diagnosed type 2 diabetes patients, aged 18 to 75 years, without neuropathy caused by other diseases or factors
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-07 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Shear Wave Velocity | from 2024-4 to 2029-4

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No